CLINICAL TRIAL: NCT05806697
Title: Investigation of AlzHeimer's Predictors in Subjective Memory Complainers - Extension Study
Acronym: INSIGHT-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C20-70
Record Dates: First submitted 2023-03-14; First posted 2023-04-10 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease; Memory Complaint; Memory Disorders
Keywords: risks factors; brain amyloid load; neurosciences; neurology; memory complaint; memory disorders
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Blood Specimen Collection; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Other)
  Interventions: Procedure: Electroencephalogram (EEG); Procedure: Oculomotor tests; Procedure: MRI; Radiation: 18-F amyloid PET Scan; Radiation: 18F-fluorodeoxyglucose (FDG) PET Scan; Biological: Blood sampling; Biological: Lumbar puncture

INTERVENTIONS:
Procedure: Electroencephalogram (EEG) — The EEG will be uniquely performed during for the whole study if a given subject converts to symptomatic AD or in the occurrence of significant cognitive decline.
Procedure: Oculomotor tests — All participants in the INSIGHT-2 study are invited to perform the oculomotor test, excepting subjects reporting oculomotor disorders.
Procedure: MRI — All INSIGHT-2 participants will undergo a baseline MRI (structural and resting state fMRI) a follow-up MRI at M12, M36 and M60.
Radiation: 18-F amyloid PET Scan — The primary endpoint is conversion to the symptomatic stage in subjects at risk, identified by positive amyloid staining (A+) on florbetapir PET imaging. Participants will receive an injection of 18F-Florbetapir prior to undergoing amyloid PET scanning. Florbetapir (18F) is an experimental imaging compound labeled with [18F] fluorine that decays by positron (β+) emission and has a half-life of 109.77 min. This procedure will be done at baseline.
Radiation: 18F-fluorodeoxyglucose (FDG) PET Scan — Participants will receive an injection of Fludeoxyglucose 18F prior to undergoing FDG-PET. The [18F]FDG is the most well-known radiopharmaceutical positron emitter, in both clinical and preclinical fields.
Biological: Blood sampling — A total of 80 ml of whole blood will be collected for each participant in the INSIGHT-2 study for routine laboratory assessment and biobank sampling.
Biological: Lumbar puncture — A lumbar puncture for cerebrospinal fluid (CSF) collection is proposed to all participants.

SUMMARY:
A regional, single-center, prospective, observational academic cohort will follow subjects who previously participated in the INSIGHT study and who agree an extension of their follow-up in the INSIGHT-2 research for additional 5-6 years. An annual multimodal evaluation (cognitive, oculomotor, biological and neuroimaging) will be proposed in order to describe the natural history of preclinical Alzheimer's disease (AD). The primary endpoint is the conversion to the symptomatic stage in subjects at risk, identified by positive amyloid staining (A+) on florbetapir positron emission tomography (PET) imaging. The size of the cohort is estimated to around 240 participants (61 A+ subjects) among the 318 participants included in the main cohort (88 A+ subjects). The follow-up in the INSIGHT-2 cohort will be lightened compared to that of the main cohort with an annual frequency of visits rather than a six-monthly one.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that previously participated in the INSIGHT cohort
* Aged 70 to 95 years old
* Having signed an informed consent
* Willing to and able undergo a baseline PET amyloid imaging
* Affiliating to the French health-care system
* Having an identified informant who has sufficient contact with the participant and has to be able to provide accurate information, at least by phone, about the participants' cognitive and functional abilities.

Exclusion Criteria:

* Clinical Dementia Rating ≥1 at screening/baseline visit only
* Fulfilling research diagnostic criteria for any type of dementia-related disorder at screening visit (clinical AD, Dementia with Lewy Bodies [DLB], fronto-temporal dementia [FTD], vascular dementia, chronic traumatic encephalopathy [CTE], Limbic-predominant Age-related TDP-43 Encephalopathy [LATE], Primary age-related tauopathy [PART)
* Presence of any medical condition associated with a long-term risk of cognitive impairment or dementia including Parkinson's disease, brain tumor, subdural hematoma, vascular malformations, territorial stroke (excluding smaller watershed strokes), chronic hydrocephalus, traumatic brain injury with neurological sequelae, active alcohol/drug abuse, major depressive disorder, schizophrenia and bipolar disorder
* Current serious or unstable illnesses (including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic or hematologic disease) that might make the subject's participation in an investigational trial unsafe
* Any contraindications for MRI/ PET scan procedure (claustrophobia, ferromagnetic object in the body), to FDG or to 18F-Florbetapir (Amyvid®).
* Hypersensitivity to the active substance or to any of the excipients of 18F-Florbetapir (Amyvid®).
* Participation in any clinical trial of an investigational product in the last 30 days before the screening (during all study duration co-inclusion in other clinical trial of an investigational product or observational research [biomarker cohort e.g.] will be possible but the information would need to be recorded).
* Unable to comply with protocol requirements in the opinion of the investigator
* Being under guardianship (safeguard of justice, curatorship or guardianship)
* Residence in skilled nursing facility, including nursing homes (EHPAD).

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2030-10-09 (Estimated); Study Completion 2030-10-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the conversion to typical AD during the 5-year follow-up. | every year through study completion, from baseline for 5 years (M60)
  Typical AD according to International Working Group (IWG) 2014 criteria = amyloid-positive participants, with an abnormal decline of episodic memory performance on the Free and Cued Selective Reminding Test

SECONDARY OUTCOMES:
Change in Clinical Dementia Rating- Sum of Boxes (CDR-SB) score compared to baseline | Each 1 year from baseline for 5 years (M60)
  CDR-SB : Hughes, Br J Psychiatry 1982; 140: 566-72
Change in different neuroimaging, biological, electrophysiological and oculomotor parameters compared to baseline | Each 1 year from baseline for 5 years (M60)
  Exploratory outcomes
Change of the score in different self-administered, informant based questionnaires (including the Quality Of Life (QOL), Ascertain Dementia 8 (AD)8 Dementia Screening Interview, Aging Brain Care Monitor) | Each 1 year from baseline for 5 years (M60)
  Exploratory outcomes
Rate of change in biomarkers measured from blood, CSF, structural and functional neuroimaging (MRI), EEG and molecular neuroimaging (18F-FDG-PET and amyloid imaging) | Each 1 year from baseline for 5 years (M60)
  Exploratory outcomes
Conversion to symptomatic non-AD cognitive disease | Each 1 year from baseline for 5 years (M60)
  Atypical AD according to IWG 2014 criteria
Diagnosis of cerebral amyloid angiopathy based on V2.0 BOSTON criteria | Each 1 year from baseline for 5 years (M60)
  As described in the following reference: Charidimou et al., Lancet Neurol. 2022 Aug;21(8):714-725

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie BOMBOIS, MD, Principal Investigator — Institut de la Mémoire et de la Maladie d'Alzheimer (IM2A)
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No